CLINICAL TRIAL: NCT02841345
Title: Characterization of Emotional Processing of Information in Bipolar Disorder and Schizophrenic Patients
Acronym: EMOBISCHI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Basic Science
Other Study IDs: 38RC11.210
Record Dates: First submitted 2016-06-16; First posted 2016-07-22 (Estimated); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Schizophrenia; Bipolar Disorder
Keywords: emotional processing; action
MeSH Terms: conditions — Schizophrenia; Bipolar Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Bipolar (Other): bipolar patients type I or II (DSM-IV TR), euthymic phase
  Interventions: Other: behavioral and fMRI
- Schizophrenic (Other): schizophrenic loss or paranoid or undifferentiated patients
  Interventions: Other: behavioral and fMRI
- Control (Other): control group (paired in age and sex for patients)
  Interventions: Other: behavioral and fMRI

INTERVENTIONS:
Other: behavioral and fMRI — The experience will include 3 sessions. Each session will consist of the presentation of a pseudo-random sequence of 24 black and white images of negative emotional natural scenes, 24 positive emotional situations and 24 neutral emotional situations.
  * In the first session, participants will carry out an emotional assessment task: it will show at the end of each test his emotional feeling - pleasant, unpleasant or nothing - using a joystick.
  * In a second session, the participant will perform a motor task decision: it will show at the end of each test the tendency to action he would handle the situation actually using 3 buttons également- approach withdrawal or neither one nor the other.
  * In the third session, the participant will perform a simple visual perception task. To be comparable to the engine plane with the other sessions, a non-categorical motor task will be requested from participants.

SUMMARY:
In the case of psychotic disorders such as bipolar disorder or schizophrenia, attention dysfunction contribute, according to the theories of neuroscience, the development of mood disorders following disturbances in the interaction-care emotion. In this context, the general objective of this research project is to refine our understanding of the similarities and distinctions between bipolar and schizophrenic patients in the basic emotional information processing. Specifically, these are: 1) to better understand what level of basic emotional information processing both conditions differ or are comparable and in what sense and 2) estimate, in both pathologies, the specific influence of the nature of the task of processing emotional information. To answer these questions, the investigators have developed a protocol to specifically target different information processing channels playing on the nature of the spatial frequency content of emotional natural scenes. To estimate in both pathologies, the specific influence of the nature of the task on emotional processing, 3 types of tasks are proposed: 1) a simple task perception and 2) -3) two tasks whose categorization one focused on the emotional feelings of the individual and the other on the tendency to action. Both tasks categorization should involve more specifically the ventromedial prefrontal cortex (CPFVM) and the dorsolateral prefrontal cortex (DLPFC) respectively. All patient data will be compared with data from healthy control participants.

DETAILED DESCRIPTION:
Main goals This research project generally aims to refine our understanding of the similarities and distinctions between bipolar and schizophrenic patients in emotional information processing.

Specifically, these are:

1. better understand what level of emotional information processing both conditions differ or are comparable and in what direction
2. assess specifically in both pathologies, emotional regulation deficits through the realization of different cognitive tasks when processing emotional information.

To answer these questions, the investigators developed an original protocol imaging functional magnetic resonance (fMRI) to specifically target different information processing channels playing on the nature of the spatial frequency content of emotional natural scenes (see Methods). emotional regulation deficits in both disorders will be addressed in part through here 3 types of tasks: 1) a simple task perception and 2) -3) two tasks categorization of which centered on the emotional feelings of the individual (task affective) and the tendency to action (motivational task). Both tasks categorization should involve more specifically the Prefrontal Cortex-Ventro Median (CPFVM) and Lateral Prefrontal Cortex-Dorso (DLPFC), respectively, distinguishing between the two categories of patients. All patient data will be compared to healthy control participants.

This project will also allow us to improve our knowledge in bipolar and schizophrenic patients compared with control subjects, i) on the brain structures of networks involved in emotional information processing and emotional regulation, ii) functional relationships still unclear between neural structures involved in both processes and iii) the nature of the information passing through these networks.

ELIGIBILITY:
healthy volunteers

Inclusion criteria

* Informed Consent signed
* Medical examination conducted before research participation
* Age, sex and level of education paired with bipolar and schizophrenic patients)
* French Language and Culture
* normal or corrected vision and hearing to normal
* affiliate Obligation to social security

Exclusion criteria

* Topic included in an ongoing experiment
* contraindication to MRI (metal hardware or electronic incompatible with MRI examination, permanent glasses, braces, Claustrophobia, cardiac or neurological stimulator, Clip unsecured vascular nonmagnetic metal Eclat)
* Important Hearing Disorders and vision
* neurological pathologies or past or current neuropsychiatric
* Family history of psychiatric disorders
* Drug treatment may modulate brain activity: benzodiazepines, antidepressants, neuroleptics, etc.
* Alcohol Ingestion
* Pregnant women, women in labor, nursing mother
* All other categories of protected persons

bipolar patients

Inclusion criteria

* Informed Consent signed
* Review medical and psychiatric assessment and inclusion made before participation in research
* Membership or beneficiary of a social security scheme
* Age over 18 years
* Language and French culture
* study BAC level or equivalent
* normal or corrected vision and hearing to normal
* Inpatient and outpatient
* Diagnosis of bipolar disorder type I and II DSM-IV TR (A.P.A 1994)
* Clinical Stability (inter-Critical) for at least three months with scores of ladders MADRS <15 and YMRS <12.
* In case of anxiety symptoms, prescription Cyanemazine® or Hydroxyzine® be allowed, at low doses (<75 mg cyamemazine and hydroxyzyne).

Exclusion criteria

* Patient Refusal
* Diagnosis of bipolar disorder with rapid cycling and mixed episodes
* psychiatric pathology addictive disorder or schizophrenia / schizoaffective
* neurological pathologies or progressive neurosurgical
* Personal history of seizures
* Treatment with electroconvulsive therapy (ECT) in the 6 months preceding the assessment.
* Patients hospitalized under stress or under legal protection measure (guardianship, curatorship)
* Subject deprived of liberty by judicial or administrative decision
* Contraindications to the practice of MRI equipment or incompatible metal or electronic foreign body with MRI examination, permanent glasses, braces, Claustrophobia, cardiac or neurological stimulator, Clip unsecured vascular nonmagnetic metal Eclat)
* significant disorders of hearing and vision
* Alcohol Ingestion
* Pregnant women, women in labor, nursing mother

schizophrenic patients

Inclusion criteria

* Informed Consent signed
* Review medical and psychiatric assessment and inclusion made before participation in research
* Membership or beneficiary of a social security scheme
* Age over 18 years
* Language and French culture
* study BAC level or equivalent
* normal or corrected vision and hearing to normal
* Inpatient and outpatient
* diagnosis of schizophrenic disorders such deficit, paranoid and undifferentiated
* clinical stability for three months with PANSS scores <120 and no mood episode characterized (MADRS <15; YMRS <12)

Exclusion criteria

* Patient Refusal
* neurological pathologies or progressive neurosurgical
* psychiatric pathology addictive
* Patients hospitalized under stress or under legal protection measure (guardianship, curatorship)
* Subject deprived of liberty by judicial or administrative decision
* Contraindications to the practice of MRI equipment or incompatible metal or electronic foreign body with MRI examination, permanent glasses, braces, Claustrophobia, cardiac or neurological stimulator, Clip unsecured vascular nonmagnetic metal Eclat)
* significant disorders of hearing and vision
* Alcohol Ingestion
* Pregnant women, women in labor, nursing mother

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2011-12; Primary Completion 2020-02-29 (Estimated); Study Completion 2020-02-29 (Estimated)

PRIMARY OUTCOMES:
Psychometric evaluation | 70 minutes
  PANSS - POSITIVE AND NEGATIVE SYNDROME SCALE Scale with 30 items
Psychometric evaluation | 15 minutes
  MADRS - Montgomery Asberg Depression Rating
Psychometric evaluation | 15 minutes
  YMRS - Young Mania Rating Scale
Self-Questionnaire | Few hours
  SHAPS - Snaith-Hamilton Pleasure Scale Starkstein STAI Y - State-Trait Anxiety Inventory AIM: "affect intensity measure" ALS: "affective lability scale" MATHYS
Cognitive questionnaire | 15 minutes
  CPT II - Conners' Continuous Performance Test II

CONTACTS AND LOCATIONS:
Overall Officials: AURELIE CAMPAGNE, PhD, Study Director — LPNC; MIRCEA POLOSAN, PhD MD Pr., Principal Investigator — GrenobleUniversityHospital
Locations (1):
- GrenobleUniversityHospital, La Tronche, France